CLINICAL TRIAL: NCT03325556
Title: A Double-blind, Placebo-controlled, Relapse Prevention Study of Pimavanserin for the Treatment of Hallucinations and Delusions Associated With Dementia-related Psychosis
Brief Title: Relapse Prevention Study of Pimavanserin in Dementia-related Psychosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-045; 2017-002227-13 (EudraCT Number)
Record Dates: First submitted 2017-10-18; First posted 2017-10-30 (Actual); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Dementia-related Psychosis
Keywords: Dementia; Dementia-related psychosis; Dementia associated with Parkinson's disease; Dementia with Lewy bodies; Alzheimer's disease; Behavioral variant frontotemporal dementia; Progressive supranuclear palsy; Corticobasal degeneration; Vascular dementia; Hallucinations; Delusions; Psychosis
MeSH Terms: conditions — Dementia; Lewy Body Disease; Alzheimer Disease; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Dementia, Vascular; Hallucinations; Delusions; Psychotic Disorders | interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Drug - Pimavanserin (Experimental)
  Interventions: Drug: Pimavanserin 34 mg; Drug: Pimavanserin 20 mg

INTERVENTIONS:
Drug: Placebo — Placebo, tablets, once daily by mouth
  Arms: Placebo
Drug: Pimavanserin 34 mg — Pimavanserin 34 mg total daily dose, tablets, once daily by mouth
  Arms: Drug - Pimavanserin
Drug: Pimavanserin 20 mg — Pimavanserin 20 mg total daily dose, tablets, once daily by mouth
  Arms: Drug - Pimavanserin

SUMMARY:
The purpose of this study is to evaluate the efficacy of pimavanserin compared to placebo in preventing relapse of psychotic symptoms in subjects with dementia-related psychosis who responded to 12 weeks of open label pimavanserin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Meets criteria for All-cause Dementia according to NIA-AA guidelines
2. Meets clinical criteria for one of the following disorders: Dementia associated with Parkinson's disease, Dementia with Lewy bodies, Possible or probable Alzheimer's disease, Frontotemporal degeneration spectrum disorders, Vascular dementia
3. Has an MMSE score ≥6 and ≤24
4. Has had psychotic symptoms for at least 2 months
5. Must be on a stable does of cholinesterase inhibitor or memantine, if applicable
6. If the subject is female, she must not be pregnant or breastfeeding. She must also be of non-childbearing potential or must agree to use a clinically acceptable method of contraception for the duration of the study

Exclusion Criteria:

1. Has psychotic symptoms that are primarily attributable to a condition other than dementia
2. Has had a recent major depressive episode
3. Has experienced suicidal ideation or behavior within 3 months prior to study enrollment
4. Has evidence of a non-neurologic medical comorbidity or medication use that could substantially impair cognition
5. Has a history of ischemic stroke within the last 12 months or any evidence of hemorrhagic stroke
6. Has a known history of cerebral amyloid angiopathy (CAA), epilepsy, CNS neoplasm, or unexplained syncope
7. Has any of the following: greater than New York Heart Association (NYHA) Class 2 congestive heart failure, Grade 2 or greater angina pectoris, sustained ventricular tachycardia, ventricular fibrillation, torsade de pointes, syncope due to an arrhythmia, an implantable cardiac defibrillator
8. Had a myocardial infarction within the last 6 months
9. Has a known personal or family history or symptoms of long QT syndrome
10. Has a significant unstable medical condition that could interfere with subject's ability to complete the study or comply with study procedures
11. Requires treatment with a medication or other substance that is prohibited by the protocol

Additional inclusion/exclusion criteria apply. Subjects will be evaluated at screening to ensure that all criteria for study participation are met.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (27):
  - ATP Clinical Research Inc., Costa Mesa, California
  - Neurology Center of North Orange County, Fullerton, California
  - Visionary Investigators Network (Aventura Neurologic Associates), Aventura, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Visionary Investigators Network (First Choice Neurology Group), Miami, Florida
  - Novel Clinical Research Center, LLC, Miami, Florida
  - Collier Neurologic Specialists LLC, Naples, Florida
  - Bioclinica Research, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Quantum Laboratories, Pompano Beach, Florida
  - Neuroscience Research Institute, Winfield, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Alzheimer Disease Center, Quincy, Massachusetts
  - Clinical Research Professionals, Chesterfield, Missouri
  - Millennium Psychiatric Associates, LLC; DBA Millennium Center for Clinical Research, St Louis, Missouri
  - Neurology Center of Las Vegas, Las Vegas, Nevada
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - BioBehavioral Health, Toms River, New Jersey
  - Neurological Associates of Albany, PC, Albany, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Abington Neurological Associates Ltd., Willow Grove, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - University of Virginia Adult Neurology, Charlottesville, Virginia
- Mental Health Center - Ruse EOOD, Rousse, Bulgaria
- Chile (3):
  - Psicomed Estudios Medicos, Antofagasta
  - Biomedica Research Group, Santiago
  - Especialidades Médicas L y S, Santiago
- Czechia (4):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Clintrial s.r.o., Prague
  - AD71, s.r.o., Prague
  - Vestra Clinics, s.r.o, Rychnov nad Kněžnou
- France (2):
  - Assistance Publique Hopitaux de Marseille (AP-HM) - Hopital de La Timone - Service de Neurologie et Pathologie du Mouvement du Pr Azulay, Marseille
  - Centre de Recherche du Gerontopole - CHU de Toulouse, Toulouse
- Klinik für Psychiatrie und Psychotherapie der Universität Tübingen, Tübingen, Germany
- Italy (5):
  - Azienda Ospedaliera di Padova Clinica Neurologica, Padua
  - IRCCS San Raffaele Pisanna, Rome
  - IRCCS Fondazione Santa Lucia, Dipartimento di Neurologia e Psichiatria, Rome
  - Universita degli Studi di ROMA "La Sapienza" Dipartimento di NEUROLOGIA E PSICHIATRIA, Rome
  - Azienda Ospedaliero-Universitaria Citta della Salute a della Scienza di Torino - c/o Presidio Ospedaliero Molinette Clinica Neurologica I, Torino
- Poland (8):
  - Przychodnia Śródmieście Sp. z o.o., Bydgoszcz
  - ISPL Wieslaw Jerzy Cubala, Gdansk
  - Care Clinic, Katowice
  - Specjalistyczna Praktyka Lekarska, Lublin
  - NZOZ Neuro-Kard Ilkowski i Partnerzy Spółka Partnerska Lekarzy, Poznan
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Siemianowice Śląskie
  - Euromedis Sp z. o. o., Szczecin
  - Centrum Medyczne NeuroProtect, Warsaw
- Serbia (8):
  - Clinical center of Serbia, Clinic for Neurology, Belgrade
  - Military Medical Academy, Clinic for Neurology, Belgrade
  - Clinical Hospital Center Dr Dragisa Misovic-Dedinje, Belgrade
  - Institut of Mental Health, Belgrade
  - Psychiatric Clinic, Military Medical Academy, Belgrade
  - Clinic for Psychiatry, Clinical Center Kragujevac, Kragujevac
  - Department of addictive disorders of the Clinic for Psychiatry, Clinical center Kragujevac, Kragujevac
  - Clinic for Psychiatry, Niš
- Slovakia (5):
  - MUDr. Beata Dupejova, neurologicka ambulancia s.r.o, Banská Bystrica
  - Epamed s.r.o., Psychiatricka ambulancia, Košice
  - NEURES s.r.o. neurologicka ambulancia, Krompachy
  - Centrum Zdravia R.B.K., s.r.o., Svidník
  - Crystal Comfort, s.r.o., Vranov nad Topľou
- Spain (5):
  - Clinica IINA, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General de Cataluña, Sant Cugat del Vallès
  - Estudio de Psiquiatría, Seville
  - Hospital Universitario Virgen del Rocío, Seville
- Ukraine (10):
  - Municipal Institution "Odesa Regional Psychiatric Hospital #2", Female Gerontological Department # 5, Male Gerontological Department #1, Oleksandrivka, Odesa Oblast
  - Communal Institution "Dnipropetrovsk Regional Clinical Hospital n.a. I. I. Mechnikov", Dnipro
  - Municipal Institution of Health Care "Kharkiv Regional Clinical Psychiatric Hospital #3", Kharkiv
  - State Institution "Institute of Neurology, Psychiatry, and Narcology of the National Academy of Medical Sciences of Ukraine", Department of Clinical, Social, and Paediatric Psychiatry, Kharkiv
  - Kherson Regional Psychiatric Hospital, Kherson
  - Lviv Regional State Clinical Psychiatric Hospital, Lviv
  - Municipal Institution "Odesa Regional Medical Center of Mental Health", Department #18, Odesa
  - Poltava Regional Clinical Psychiatric Hospital named after O.F. Maltsev, Poltava
  - Municipal Institution "Vinnytsya Regional Psychoneurological Hospital n.a. Acad. O.I.Yushchenko", Male Department #14, Female Department #15, Vinnytsya National Medical University n.a. M.I.Pyrogov, Department of Psychiatry, Narcology and Psychotherapeutic, Vinnytsia
  - Municipal Institution "Zaporizhzhya Regional Clinical Hospital of Zaporizhzhya Regional Council", Zaporizhzhya
- United Kingdom (4):
  - Royal United Hospital - The Research Institute for the Care of Older People (RICE) Centre, Bath
  - MAC Clinical Research - Blackpool, Blackpool
  - Re:Cognition Health Ltd., London
  - MAC Clinical Research - Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torres-Yaghi Y, Chrones L, Abler V, Brunson G. Safety and efficacy of pimavanserin in patients with Lewy body dementia experiencing dementia-related psychosis in the HARMONY study. BMC Neurol. 2025 Nov 24;25(1):479. doi: 10.1186/s12883-025-04496-8. PMID 41286676
- [Derived] Cummings JL, Ismail Z, Dickerson BC, Ballard C, Grossberg G, McEvoy B, Foff E, Atri A. Development and assessment of a brief screening tool for psychosis in dementia. Alzheimers Dement (Amst). 2021 Dec 7;13(1):e12254. doi: 10.1002/dad2.12254. eCollection 2021. PMID 34934801
- [Derived] Tariot PN, Cummings JL, Soto-Martin ME, Ballard C, Erten-Lyons D, Sultzer DL, Devanand DP, Weintraub D, McEvoy B, Youakim JM, Stankovic S, Foff EP. Trial of Pimavanserin in Dementia-Related Psychosis. N Engl J Med. 2021 Jul 22;385(4):309-319. doi: 10.1056/NEJMoa2034634. PMID 34289275
- See also: Tariot P, et al. HARMONY relapse-prevention study: pimavanserin significantly prolongs time to relapse of dementia-related psychosis. J Prev Alz Dis. 2019; 6(suppl 1):S30-S31 — https://link.springer.com/article/10.14283/jpad.2019.47

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed in subjects with all-cause dementia according to NIA-AA guidelines, including dementia associated with Parkinson's disease, dementia with Lewy Bodies, possible or probable Alzheimer's disease, frontotemporal degeneration spectrum disorder, and/or vascular dementia, and were to have had at least a 2-month history of psychotic symptoms.
Pre-assignment Details: During the screening period, subjects were assessed for study eligibility and prohibited medications were discontinued when medically appropriate. Subjects and partner/caregivers also received a standardized psychosocial therapy training.
Groups:
- Pimavanserin Open-Label Period: Pimavanserin 34 mg once daily, with the possibility to adjust to pimavanserin 20 mg once daily between Weeks 1 and 4 based on tolerability. After Week 4, the dose of study drug remained fixed at either 34 or 20 mg once daily.
- Pimavanserin Double-Blind Period: Pimavanserin 34 mg once daily or pimavanserin 20 mg once daily (the dose at which patients completed the Open-Label Period) for 26 weeks or until relapse
- Placebo Double-Blind Period: Placebo once daily for 26 weeks or until relapse
Period: Open-label Period
Arm/Group | Pimavanserin Open-Label Period | Pimavanserin Double-Blind Period | Placebo Double-Blind Period
Started | 392 | 0 | 0
Completed | 217 | 0 | 0
Not Completed | 175 | 0 | 0
Not completed — Lack of Response in OL period | 70 | 0 | 0
Not completed — Adverse Event | 27 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Non-compliance with study drug | 5 | 0 | 0
Not completed — Use of prohibited medication | 1 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 0 | 0
Not completed — Not otherwise specified | 8 | 0 | 0
Not completed — Administrative discont. at study termination | 41 | 0 | 0
Period: Double-blind Period
Arm/Group | Pimavanserin Open-Label Period | Pimavanserin Double-Blind Period | Placebo Double-Blind Period
Started | 0 | 105 | 112
Completed | 0 | 44 | 35
Not Completed | 0 | 61 | 77
Not completed — Relapse | 0 | 15 | 34
Not completed — Adverse Event | 0 | 3 | 1
Not completed — Noncompliance with study drug | 0 | 0 | 1
Not completed — Use of prohibited medication | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 6 | 4
Not completed — Not otherwise specified | 0 | 1 | 5
Not completed — Administrative discont. at study termination | 0 | 35 | 31

BASELINE CHARACTERISTICS:
Population: Patients who entered the respective study period and received at least one dose of study medication
Arm/Group | Pimavanserin Open-Label Period
Number analyzed (Participants) | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229
  Male | 163
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: For 8 patients, Information on race was not available.
  Participants
    number analyzed (Participants) | 384
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 10
    White | 371
    More than one race | 0
    Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 118
  Czechia | 11
  Ukraine | 74
  United Kingdom | 8
  Spain | 9
  Poland | 42
  Italy | 13
  Slovakia | 35
  Bulgaria | 3
  Chile | 27
  France | 7
  Serbia | 44
  Germany | 1
Dementia severity [Count of Participants; unit: Participants]
  Mild | 65
  Moderate | 275
  Severe | 52
Scale for the Assessment of Positive Symptoms-Hallucinations+Delusions (SAPS-H+D) total score [Mean (Standard Deviation); unit: Score on a scale] — The Scale for the Assessment of Positive Symptoms-Hallucinations and Delusions (SAPS-H+D) is a 20-item scale; the total score is the sum of the 20 item scores (range 0-100); higher scores denote more severe symptoms.
  Score on a scale | 24.4 (9.22)
Clinical Global Impression-Severity (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression-Severity (CGI-S) is a clinician-rated, 7-point scale to rate the severity of the patient's hallucinations and delusions at the time of assessment. Scores range from 1 to 7, with a higher score marking a more severe state.
  units on a scale | 4.7 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Relapse in the Double-blind (DB) Period
Description: The time from randomization to relapse in the DB period was compared between treatment groups using a Cox regression model. The treatment effect was measured by the hazard ratio (HR).
  Relapse was defined as (1) ≥30% increase in SAPS-H+D total score from DB baseline (BL) and CGI-I score ≥6 relative to DB BL, (2) treatment with antipsychotic for dementia-related delusions/hallucinations, (3) treatment/study discontinuation due to lack of efficacy, and/or (4) hospitalization for worsening dementia-related psychosis.
  SAPS-H+D is a 20-item scale; the total score is the sum of the 20 item scores (range 0-100); higher scores denote more severe symptoms. CGI-I is a clinician-rated 7-point scale to rate improvement in hallucinations/delusions relative to BL (range 1-7); higher scores denote less improvement or worsening.
  A pre-specified IA was conducted after accrual of 40 adjudicated relapse events. The prespecified stopping criterion was met; the study was stopped for efficacy.
Time Frame: From randomization in the DB period through 26 weeks
Population: All patients randomized on or before the database cutoff date for the IA (i.e., when 40 adjudicated relapse events had accrued).
Measure: Median (Full Range); unit: days
Arm/Group | Pimavanserin Double-Blind Period | Placebo Double-Blind Period
Number analyzed (Participants) | 95 | 99
days | NA [NA to NA] — The median time to relapse could not be estimated as the Kaplan-Meier probability estimate of relapse over the 26-week DB period did not exceed 50%. | NA [NA to NA] — The median time to relapse could not be estimated as the Kaplan-Meier probability estimate of relapse over the 26-week DB period did not exceed 50%.
Statistical Analysis 1: Comparison: Pimavanserin Double-Blind Period vs Placebo Double-Blind Period; Test type: Superiority; p = 0.0023, Regression, Cox — 1-sided p-value reported. The protocol-defined O'Brien Flemming stopping boundary for the planned IA was a 1-sided p-value equal to 0.0033; Hazard Ratio (HR) = 0.353, 95% CI 2-sided [0.172 to 0.727], Standard Error of Mean 0.3676 — Model included covariates for Treatment group, dementia subtype, and region, and robust sandwich-type variance estimator

2. Secondary Outcome: Time From Randomization to Discontinuation From the DB Period for Any Reason
Description: The endpoint of time from randomization to discontinuation from the DB period for any reason (other than termination of the study by the sponsor) was compared between treatment groups using a Cox regression model. The treatment effect was measured by the HR.
Time Frame: From randomization in the DB period through 26 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Pimavanserin Double-Blind Period | Placebo Double-Blind Period
Number analyzed (Participants) | 95 | 99
days | NA [NA to NA] — The median time to discontinuation could not be estimated as the Kaplan-Meier probability estimate over the 26-week DB period did not exceed 50%. | NA [NA to NA] — The median time to discontinuation could not be estimated as the Kaplan-Meier probability estimate over the 26-week DB period did not exceed 50%.
Statistical Analysis 1: Comparison: Pimavanserin Double-Blind Period vs Placebo Double-Blind Period; Test type: Superiority; p = 0.0024, Regression, Cox — 1-sided p-value; Hazard Ratio (HR) = 0.452, 95% CI 2-sided [0.261 to 0.785], Standard Error of Mean 0.2812 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were to be documented through 30 days after the last dose in the study.
Arm/Group | Pimavanserin Open-Label Period | Pimavanserin Double-Blind Period | Placebo Double-Blind Period
All-Cause Mortality (participants affected / at risk) | 1/392 | 1/105 | 0/112
Serious Adverse Events (participants affected / at risk) | 20/392 | 5/105 | 4/112
Other Adverse Events (participants affected / at risk) | 24/392 | 16/105 | 9/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin Open-Label Period (N=392) | Pimavanserin Double-Blind Period (N=105) | Placebo Double-Blind Period (N=112)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic encephalopathy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Agression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropsychiatric symptoms (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin Open-Label Period (N=392) | Pimavanserin Double-Blind Period (N=105) | Placebo Double-Blind Period (N=112)
Urinary tract infection (Infections and infestations) | 18 (19) | 6 (8) | 4 (5)
Headache (Nervous system disorders) | 6 (6) | 10 (13) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT03325556/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT03325556/SAP_001.pdf